CLINICAL TRIAL: NCT05236218
Title: Patients' Treatment Preferences For Muscle Invasive Bladder Cancer Cancer: A Discrete Choice Experiment
Brief Title: To Better Understand the Most Important Factors for Patients When They Decide on the Type of Treatment They Receive for Muscle Invasive Bladder Cancer (MIBC).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: PTPDCE
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Muscle Invasive Bladder Cancer; Surgery; Sexual Wellbeing; Patient Satisfaction; Patient Preference
Keywords: Muscle invasive bladder cancer; Patient Preference
MeSH Terms: conditions — Patient Satisfaction; Patient Preference | interventions — delta 24-sterol reductase; Pilot Projects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilot study (n = 10): 10 participants will be recruited to complete the questionnaire (version 1). A research assistant will be present to help support them /answer any questions around the format. Readability and comprehension will be noted. Any changes (if needed) can be implemented to its format before the main data collection.
  Interventions: Other: Semi-Structured Interview Patients Interview
- Discrete Choice Experiment Questionnaire (n = 50): Discrete Choice Experiment (DCE) Patients
  Interventions: Other: Discrete Choice Experiment (DCE) Patients DCE Questionnaire

INTERVENTIONS:
Other: Discrete Choice Experiment (DCE) Patients DCE Questionnaire — Discrete Choice Experiment (DCE) Patients
  Groups: Discrete Choice Experiment Questionnaire (n = 50)
Other: Semi-Structured Interview Patients Interview — First version of questionnaire (readability/comprehension check)
  Other Names: Pilot study
  Groups: Pilot study (n = 10)

SUMMARY:
Through our study, we aim to understand the most important factors for patients when they decide on the type of treatment they receive for MIBC. Our study consists of a discrete choice experiment (DCE): a type of questionnaire used to elicit preferences in the absence of data. DCEs are frequently used in oncological research to elicit preferences from participants without directly asking them to state their preferred options. Participants undertaking our DCE questionnaire will presented with a series of alternative hypothetical scenarios containing several variables or "attributes" (5), each of which may have a number of variations or "levels".

DETAILED DESCRIPTION:
The study will be conducted using validated and established protocols for undertaking DCEs. A literature review was undertaken to assess what the most important considerations where for patients when making decisions about the treatment they receive for MIBC. Using this literature search as a starting point, discussion groups with relevant healthcare professionals and service users were undertaken to decide on the final attribute and levels for the questions. Five attributes were selected through an iterative process - Body image, Life expectancy, Side-effects from treatment, Living as bladder cancer survivor, and Sexual wellbeing

The study is divided into three stages:

1. Interviews with experienced healthcare professionals and service users to finalise attributes and levels to be used for the questionnaire
2. A representative sample of patients (~10) will be asked to complete the questionnaire in addition to a brief unstructured interview to assess understanding (e.g. readability and ease of completing the questionnaire)
3. Necessary changes based on feedback from the pilot study will be applied before the main study is carried out

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MIBC cancer and currently undergoing treatment or have previously completed treatment for MIBC

Exclusion Criteria:

* Any of other type of bladder cancer (unknown, metastatic, or non muscle invasive bladder cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women with diagnosed MIBC who are currently undergoing treatment or have previously completed treatment for MIBC
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-04-25 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Willingness to accept treatment attributes, and trade-offs between these, using a study-specific Discrete Choice Experiment (DCE) Questionnaire | Through study completion, an average of 1 year (Discrete Choice Experiment (DCE) Questionnaire). Trade-off from Marginal Rate of Substitution calculate as percentage points (0 to 100). ]

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hughes, Principal Investigator — KCL/GSTTH
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided